CLINICAL TRIAL: NCT02345460
Title: Preoperative Folfirinox for Resectable Pancreatic Adenocarcinoma - A Phase II Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Competing studies
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE4214; NCI-2014-02277 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE4214 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2015-01-20; First posted 2015-01-26 (Estimated); Results first posted 2018-07-13 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-06

CONDITIONS: Pancreatic Adenocarcinoma; Poorly Differentiated Malignant Neoplasm; Resectable Pancreatic Cancer; Stage IA Pancreatic Cancer; Stage IB Pancreatic Cancer; Stage IIA Pancreatic Cancer; Stage IIB Pancreatic Cancer; Stage III Pancreatic Cancer; Undifferentiated Pancreatic Carcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Irinotecan; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (FOLFIRINOX) (Experimental): Patients receive FOLFIRINOX regimen comprising irinotecan hydrochloride IV over 90 minutes, oxaliplatin IV over 120 minutes, leucovorin calcium IV over 120 minutes, and fluorouracil IV over 1-2 minutes and then continuously over 46 hours on day 1. Treatment repeats every 14 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Irinotecan Hydrochloride; Drug: Oxaliplatin; Drug: Leucovorin Calcium; Drug: Fluorouracil; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Irinotecan Hydrochloride — Given IV
Drug: Oxaliplatin — Given IV
Drug: Leucovorin Calcium — Given IV
  Other Names: CF
Drug: Fluorouracil — Given IV
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well combination chemotherapy works in treating patients with pancreatic cancer before undergoing surgery. Drugs used in chemotherapy, such as irinotecan hydrochloride, oxaliplatin, leucovorin calcium, and fluorouracil (FOLFIRINOX), work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving more than one drug (combination chemotherapy) before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine feasibility of preoperative FOLFIRINOX for resectable pancreatic adenocarcinoma.

SECONDARY OBJECTIVES:

I. To determine safety and toxicity of preoperative FOLFIRINOX. II. To determine response rate. III. To determine proportion achieving major pathologic response - per College of American Pathologists (CAP) criteria.

IV. To determine proportion achieving R0 resection. V. To determine perioperative (30-day) mortality. VI. To determine the role of cancer antigen (CA)19.9 as potential prognostic and/or predictive biomarker.

VII. To determine progression-free survival. VIII. To determine overall survival.

OUTLINE:

Patients receive FOLFIRINOX regimen comprising irinotecan hydrochloride intravenously (IV) over 90 minutes, oxaliplatin IV over 120 minutes, leucovorin calcium IV over 120 minutes, and fluorouracil IV over 1-2 minutes and then continuously over 46 hours on day 1. Treatment repeats every 14 days for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed carcinoma of the pancreas; most cases will be adenocarcinoma; cases with "undifferentiated" or "poorly differentiated" carcinoma will also be eligible
* There should be no evidence of metastatic disease on imaging of the chest, abdomen, and pelvis; this imaging should be either a contrast-enhanced computed tomography (CT) scan, or a contrast-enhanced magnetic resonance imaging (MRI) scan; positron emission tomography (PET) scans alone will not be adequate alternatives; there should be no evidence of occult metastatic disease in the abdomen, confirmed by laparoscopic examination
* The primary tumor must be resectable, defined as no involvement (abutment or encasement) of the major arteries (celiac, common hepatic, superior mesenteric) and interface between tumor and vessel (portal, superior mesenteric veins) wall to be less than 180 degrees of the circumference of the vessel wall; this should be confirmed by imaging of the abdomen, either by a contrast-enhanced computed tomography (CT) scan, or a contrast-enhanced magnetic resonance imaging (MRI) scan; PET scans will not be adequate alternatives; for each patient, the resectability must be reviewed by one of the study surgeons
* Patient must not have received any cancer-directed therapy (e.g., surgery, chemotherapy, radiation therapy, biologic therapy) for the index diagnosis
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Hemoglobin >= 10.0 g/dl
* Absolute neutrophil count >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Total bilirubin =< 1.5 X institutional upper limit of normal
* Serum creatinine within normal institutional limits, or creatinine clearance (calculated by Cockcroft-Gault) >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Women of child-bearing potential and men must agree to use adequate contraception (double-barrier method of birth control or abstinence) for the duration of study participation and for 6 months after completing chemotherapy; should a woman become pregnant or suspect that she is pregnant while she or her partner is participating in this study, she should inform the treating physician immediately
* Subjects must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or breastfeeding women
* Pre-existing peripheral neuropathy (grade I or higher)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-09; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Davendra Sohal, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (FOLFIRINOX)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (FOLFIRINOX)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Undergoing Surgical Resection After Receiving at Least 4 of the 6 Courses of Preoperative Chemotherapy
Description: Proportion will be estimated using a binomial test.
Time Frame: Up to 12 weeks
Population: Only 1 patient was enrolled on study. Outcome data was not analyzed. Trial closed due to competing studies.
Arm/Group | Treatment (FOLFIRINOX)
Number analyzed (Participants) | 0

2. Secondary Outcome: Progression-free Survival
Description: Time from enrollment to the earlier of death or disease progression. Will be estimated with Kaplan Meier curves.
Time Frame: Up to 2 years
Population: Only 1 patient was enrolled on study. Outcome data was not analyzed. Trial closed due to competing studies.
Arm/Group | Treatment (FOLFIRINOX)
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival
Description: Time from enrollment to death from any cause. Will be estimated with Kaplan Meier curves.
Time Frame: Up to 2 years
Population: Only 1 patient was enrolled on study. Outcome data was not analyzed.
Arm/Group | Treatment (FOLFIRINOX)
Number analyzed (Participants) | 0

4. Secondary Outcome: Incidence of Toxicities Greater Than Grade 2, Using the Common Terminology Criteria for Adverse Events Version 4.0
Description: Toxicity evaluation will be enumeration of all major toxicities, with proportions calculated for each.
Time Frame: Up to 30 days after end of treatment or to the day prior to surgery
Population: Only 1 patient was enrolled on study. Outcome data was not analyzed. Trial closed due to competing studies.
Arm/Group | Treatment (FOLFIRINOX)
Number analyzed (Participants) | 0

5. Secondary Outcome: Response Rate Assessed Using Response Evaluation Criteria in Solid Tumors Version 1.1
Description: Will be calculated as a binary outcome. Exact 95% confidence intervals will be calculated for binary outcomes.
Time Frame: Up to 2 years
Population: Only 1 patient was enrolled on study. Outcome data was not analyzed. Trial closed due to competing studies.
Arm/Group | Treatment (FOLFIRINOX)
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Participants Achieving Major Pathologic Response
Description: Will be calculated as a binary outcome. Exact 95% confidence intervals will be calculated for binary outcomes.
Time Frame: Up to 2 years
Population: Only 1 patient was enrolled on study. Outcome data was not analyzed. Trial closed due to competing studies.
Arm/Group | Treatment (FOLFIRINOX)
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants Achieving R0 Resection
Description: Will be calculated as a binary outcome. Exact 95% confidence intervals will be calculated for binary outcomes.
Time Frame: Up to 2 years
Population: Only 1 patient was enrolled on study. Outcome data was not analyzed. Trial closed due to competing studies.
Arm/Group | Treatment (FOLFIRINOX)
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Participants Experiencing Perioperative (30-day) Mortality
Description: Will be calculated as a binary outcome. Exact 95% confidence intervals will be calculated for binary outcomes.
Time Frame: Up to 30 days
Population: Only 1 patient was enrolled on study. Outcome data was not analyzed. Trial closed due to competing studies.
Arm/Group | Treatment (FOLFIRINOX)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Treatment (FOLFIRINOX)
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes